CLINICAL TRIAL: NCT05646771
Title: Feasibility Study for Collaborate2Lose: Collaborating With Support Persons to Improve Long-term Weight Loss
Brief Title: Feasibility Study for Collaborate2Lose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: William S. Middleton Memorial Veterans Hospital (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0629; SMPH/SURGERY/WISOR (Other: UW Madison); Protocol Version 1/24/23 (Other: UW Madison)
Record Dates: First submitted 2022-12-02; First posted 2022-12-12 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: All participants will receive the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Partner-Supported (Experimental): Dyads comprised of one Veteran and a cohabitating support person will participate in a behavioral weight management intervention.
  Interventions: Behavioral: Partner support

INTERVENTIONS:
Behavioral: Partner support — Remotely delivered, partner-supported weight management counseling delivered in group visits every two weeks over 14 weeks (8 sessions)

SUMMARY:
In this feasibility study, dyads comprising a Veteran with obesity and a cohabiting adult support person will participate in group-based weight management counseling. Counseling will be delivered using an approved virtual technology platform. The curriculum is based on the VA national MOVE! weight management curriculum and involves additional content focusing on couples' communication skills.

ELIGIBILITY:
Inclusion Criteria (Veteran):

1. Aged 18 years or older
2. BMI ≥ 30 kg/m2
3. Had at least one visit with their primary care provider at the Madison VA within the past year (in-person or telehealth)
4. Weight ≤ 420lbs due to limit of the study scales
5. Cohabitating and daily contact for at least the past 6 months with an adult who can provide support (e.g. spouse/domestic partner, sibling, friend, family member) during the study period
6. Desire to lose weight
7. Ability to speak English
8. Agrees to attend visits per protocol
9. Score of at least 4 out of 6 on a validated cognitive screener
10. Access to hardware and internet connection to enable participation with approved virtual platform
11. Individual email address
12. Able to stand on a scale without assistance

Exclusion Criteria (Veteran):

1. Medication other than metformin, incretin mimetics and incretin enhancers for type 2 diabetes due to increased risk for hypoglycemia
2. Active dementia, psychiatric illness, or substance abuse
3. History of bariatric surgery
4. Diuretic medication doses higher than hydrochlorothiazide 25 mg daily, furosemide 40 mg daily, Torsemide 20 mg daily, Bumetanide 1 mg daily or any use of Metolazone). Use of potassium-sparing diuretics is acceptable.
5. Chronic kidney disease at stage 4 or higher
6. Participation in MOVE! in the past 3 months
7. Currently enrolled in a research or clinical program focusing on lifestyle change
8. Pregnancy or planning to become pregnant in the next 18 months, or breastfeeding
9. Psychiatric illness not well-controlled by medication or therapy
10. Score ≥ 8 on alcohol abuse screener
11. Use of any drugs not prescribed, excluding cannabis
12. Weight loss ≥ 10lb in the month prior to screening
13. Living in a facility such as a nursing home, skilled nursing facility, or assisted living facility
14. Is unable to control what food is prepared and/or served in household
15. Problems with hearing that prevent attendance to a virtual class and talking on the telephone
16. Currently enrolled in a research or clinical program focusing on lifestyle change
17. History of bariatric surgery (reconfirm) or planning to have bariatric surgery in the next 18 months
18. Current use of weight loss medications
19. Worsening heart failure requiring medication dose change in the past 6 months
20. Hospitalization for heart problems in the past 6 months
21. Current treatment or treatment in the past 6 months for cancer (besides non-melanoma skin cancers)
22. Dizziness or lightheadedness at rest or associated with physical activity
23. Chest pain in the past 6 months

Inclusion Criteria (support person):

1. Aged 18 years or older
2. Willing to participate
3. Score of at least 4 out of 6 on a validated cognitive screener
4. Ability to speak English

Exclusion Criteria (support person):

1. Underweight (BMI < 18.5 kg/m2)
2. Active dementia, uncontrolled psychiatric illness, or substance abuse
3. Living in a facility such as a nursing home, skilled nursing facility, or assisted living facility
4. Problems with hearing that prevent attendance to a virtual class and talking on the telephone
5. Any severe health issue that would impair the partner's ability to provide support

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-03-13 (Actual); Primary Completion 2023-08-08 (Actual); Study Completion 2023-08-08 (Actual)

PRIMARY OUTCOMES:
Screening to enrollment ratio | baseline
  We will calculate the screening to enrollment ratio. Our feasibility metric is 2:1 (i.e., 2 people start the phone screening in order to have one provide consent).
Retention Rate for primary outcome | 16 weeks
  The outcome assessment retention rate at 16 weeks will be calculated as [#of index participants who provide a weight at 16 weeks/number who provided a baseline weight]. Our metric is at least 80% retention at 16 weeks.

SECONDARY OUTCOMES:
Weight | 16 weeks
  Weight at 16 weeks is the primary endpoint. Veterans will be asked to weigh themselves during a virtual study visit, on a study-provided scale, while wearing light clothing (i.e., no outerwear such as jackets), with shoes removed.
Intervention adherence | 14 weeks
  Intervention adherence is calculated as the average number of group sessions attended by index participants.

CONTACTS AND LOCATIONS:
Overall Officials: Corrine Voils, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No